CLINICAL TRIAL: NCT02192944
Title: Comparison of the Electrocardiographic Effects in Relation to Pharmacokinetic Profile of Chloroquine and Piperaquine in Healthy Thai Subjects
Brief Title: Comparison of the ECG Effects Related to Pharmacokinetic Profile of Chloroquine and Piperaquine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FTM1401
Record Dates: First submitted 2014-07-01; First posted 2014-07-17 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: ECG; Pharmacokinetic profile
MeSH Terms: interventions — Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chloroquine (Active Comparator): Chloroquine base 600 mg single dose
  Interventions: Drug: Dihydroartemisinin-piperaquine
- Dihydroartemisinin-piperaquine (Active Comparator): Dihydroartemisinin-piperaquine 120/960 mg single dose
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: Chloroquine — Chloroquine base 600 mg single dose. To monitor ECG 12 lead at 0 (pre-dose), 1, 2, 4, 8, 12 and 24 hours after dosing.
  Arms: Dihydroartemisinin-piperaquine
Drug: Dihydroartemisinin-piperaquine — Dihydroartemisinin-piperaquine 120/960 mg single dose To monitor ECG 12 lead at: 0 (pre-dose), 1, 2, 4, 8, 12 and 24 hours after dosing.
  Arms: Chloroquine

SUMMARY:
Chloroquine and piperaquine are the two most widely used antimalarial drugs ever. Hundreds of millions of people have received these drugs. Both are structurally similar and have cardiovascular effect. While there are no concerns over the use of chloroquine, regulatory authorities have suggested restrictions on the use of piperaquine.

We have recently completed a series of cross-over clinical and pharmacokinetic evaluations of chloroquine, piperaquine, pyronaridine and primaquine in healthy subjects. These studied were approved by the ethical committee of FTM. All drugs were well tolerated with no clinically significant ECG changes. Four subjects were in two studies. This offers a unique opportunity to compare the electrocardiographic effects of chloroquine and piperaquine in the same subjects and therefore characterize the concentration-effect relationships, and thus relative safety.

We propose to extend the previous subject study to recruit 16 subjects including those who have received either piperaquine or chloroquine in our previous studies so that 20 subjects received both drugs for a crossover comparison. The blood sampling schedule and electrocardiograms would be exactly the same as previously but would finish at 24 hours.

DETAILED DESCRIPTION:
The investigator team has recently completed two cross-over clinical and pharmacokinetic evaluations chloroquine and piperaquine in healthy subjects i.e. Study A and Study B.

Study A: Phase 1, Open-Label Study to Evaluate Potential Pharmacokinetic Interaction of Orally Administered Primaquine and Chloroquine in Healthy Thai Adult Subjects

Study B: Open-Label Study to Evaluate Potential Pharmacokinetic Interaction of Orally Administered Primaquine and Dihydroartemisinin-Piperaquine in Healthy Adult Subjects

Four subjects were in both studies. The investigator proposes to extend the previous subject study to recruit 16 subjects including but not limited to those who have received either chloroquine from study A or piperaquine form study B in our previous studies so that 20 subjects received both drugs for a crossover comparison.

Subjects who were previously enrolled into study A that received a single dose of 600 mg chloroquine base will receive a single dose of piperaquine phosphate (in form of 120/960 mg dihydroartemisinin-piperaquine) in this study. The subjects who were previously enrolled into study B that received a single dose of piperaquine phosphate (in form of 120/960 mg dihydroartemisinin-piperaquine) will receive a single dose of 600 mg of chloroquine base in this study.

The investigator team may recruit naive subject in case, the team can't reach total number of 20 subjects.

The total duration for each subject's participation in the study is approximately 3 weeks for subject who challenges only one study drug or 11 weeks for subject who challenges both drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as judged by a responsible physician with no abnormality identified on a medical evaluation including medical history and physical examination
2. Male and female subjects aged between 18 years to 60 years.
3. A female is eligible to enter and participate in this study if she is:

   * of non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy
   * or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle stimulating hormone levels >40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy
   * or of childbearing potential, has a negative serum pregnancy test at screening and prior to start the study drug in each period, and abstain from sexual intercourse or agrees to using effective contraceptive methods (e.g., intrauterine device, hormonal contraceptive drug, tubal ligation or female barrier method with spermicide) until study completion.
4. A male is eligible to enter and participate in this study if he: agrees to abstain from (or use a condom during) sexual intercourse with females of childbearing potential or lactating females; or is willing to use a condom/spermicide, until study completion.
5. Normal electrocardiogram (ECG) with QTc < 450 msec.
6. Provide a signed and dated written informed consent prior to study participation.

Exclusion Criteria:

1. Females who are pregnant, trying to get pregnant, or are lactating.
2. The subject has evidence of active substance abuse that may compromise safety, pharmacokinetics, or ability to adhere with protocol instructions.
3. A positive pre-study hepatitis B surface antigen, positive hepatitis C antibody, or positive human immunodeficiency virus-1 (HIV-1) antibody result at screening.
4. Subjects with a personal history of hypertension, cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for torsades de points (heart failure, hypokalemia).
5. Subjects with a family history of sudden cardiac death.
6. A creatinine clearance <70 mL/min as determined by Cockcroft-Gault equation:

   CLcr (mL/min) = (140 - age) * Wt / (72 * Scr) (multiply answer by 0.85 for females) Where age is in years, weight (wt) is in kg, and serum creatinine (Scr) is in units of mg/dL [Cockcroft, 1976].
7. History of alcohol or substance abuse or dependence within 6 months of the study: History of regular alcohol consumption averaging >7 drinks/wk for women or >14 drinks/wk for men. One drink is equivalent to 12 g alcohol = 5 oz (150 mL) of wine or 12 oz (360 mL) of beer or 1.5 oz (45 mL) of 80 proof distilled spirits within 6 months of screening.
8. Use of prescription or non-prescription drugs except paracetamol at doses of up to 2 grams/day, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication until the completion of the follow-up procedure, unless in the opinion of investigator, the medication will not interfere with the study procedures or compromise subject safety.
9. The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of study medication.
10. The subject is unwilling to abstain from ingesting alcohol within 48 hours prior to the first dose of study medication until collection of the final pharmacokinetic sample.
11. Subjects who have donated blood to the extent that participation in the study would result in more than 300 mL blood donated within a 30-day period. Note: This does not include plasma donation.
12. Subjects who have a history of allergy to the study drug or drugs of this class, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates participation in the trial. In addition, if heparin is used during pharmacokinetic sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
13. Those who, in the opinion of the investigator, have a risk of non-compliance with study procedures.
14. AST or ALT >1.5 upper limit of normal (ULN).
15. Subjects with history of renal disease, hepatic disease, and/or cholecystectomy.
16. Abnormal methaemoglobin level.
17. Subjects who have anemia, Hb <12 for both male and female
18. History of antimalarial drugs use within 12 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Changes of QTc within 24 hours after dosing | 24 hours after dosing
Area under the curve | 24 hours after dosing
  Area under the curve within 24 hours after dosing

SECONDARY OUTCOMES:
Number of participant with adverse event | 24 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Borimas Hanboonkunupakarn, MD, Principal Investigator — Faculty of Tropical Medicine, Mahidol University, Thailand
Locations (1):
- Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand